CLINICAL TRIAL: NCT04471428
Title: A Phase III, Multicenter, Randomized, Open-Label, Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Atezolizumab Given in Combination With Cabozantinib Versus Docetaxel Monotherapy in Patients With Metastatic Non-Small Lung Cancer Previously Treated With an Anti-PD-L1/PD-1 Antibody and Platinum-Containing Chemotherapy
Brief Title: Study of Atezolizumab in Combination With Cabozantinib Versus Docetaxel in Patients With Metastatic Non-Small Cell Lung Cancer Previously Treated With an Anti-PD-L1/PD-1 Antibody and Platinum-Containing Chemotherapy
Acronym: CONTACT-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41892
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib; atezolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Cabozantinib (Experimental): Participants received atezolizumab on Day 1 of each 21-day cycle and cabozantinib orally once daily on Days 1-21 of each cycle.
  Interventions: Drug: Cabozantinib; Drug: Atezolizumab
- Docetaxel (Active Comparator): Participants received docetaxel on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be administered orally, once daily at a dose of 40 mg on Days 1-21 of each cycle.
  Arms: Atezolizumab + Cabozantinib
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Atezolizumab + Cabozantinib
Drug: Docetaxel — Docetaxel will be administered by IV infusion at a starting dose of 75mg/m2 on Day 1 of each 21-day cycle.
  Arms: Docetaxel

SUMMARY:
This is a Phase III, multicenter, randomized, open-label study designed to evaluate the efficacy, safety, and pharmacokinetics of atezolizumab given in combination with cabozantinib compared with docetaxel monotherapy in patients with metastatic NSCLC, with no sensitizing EGFR mutation or ALK translocation, who have progressed following treatment with platinum-containing chemotherapy and anti-PD-L1/PD-1 antibody, administered concurrently or sequentially.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic NSCLC
* Documented radiographic disease progression during or following treatment with platinum-containing chemotherapy and anti-PD-L1/PD-1 antibody, administered concurrently or sequentially for metastatic NSCLC
* Measurable disease per RECIST v1.1 outside CNS as assessed by investigator
* Known PD-L1 status or availability of tumor tissue for central PD-L1 testing
* ECOG Performance Status score of 0 or 1
* Recovery to baseline or Grade <=1 NCI CTCAE v5.0 from toxicities related to any prior treatments, unless adverse events are clinically nonsignificant and/or stable on supportive therapy in the opinion of the investigator
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs,
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm.

Exclusion Criteria:

* Prior therapy with the following agents for NSCLC: Cabozantinib, Docetaxel, Combination of an anti-PD-L1/PD-1 antibody concurrently with a vascular endothelial growth factor (VEGF)R targeting tyrosine kinase inhibitor (TKI)
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Documentation of known sensitizing mutation in the EGFR gene or ALK fusion oncogene
* Patients with known ROS1 rearrangements, BRAF V600E mutations, or other actionable oncogenes with approved therapies if available
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (more frequently than once monthly)
* Severe hepatic impairment
* Uncontrolled or symptomatic hypercalcemia
* Any other active malignancy at the time of initiation of study treatment or diagnosis of another malignancy within 3 years prior to initiation of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, incidental prostate cancer, or carcinoma in situ of the prostate, cervix, or breast
* Stroke, transient ischemic attack, myocardial infarction or other symptomatic ischemic events within 6 months of initiation of study treatment
* Significant vascular disease within 6 months of initiation of study treatment
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion on the investigator, could impact patient safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Current treatment with anti-viral therapy for HBV
* Major surgical procedure, other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Pregnant or lactating females, or intention of becoming pregnant during the treatment with atezolizumab in combination with cabozantinib in the experimental arm or during the treatment with docetaxel in the control arm, or within 5 months after the final dose of atezolizumab and/or 4 months after the final dose of cabozantinib, whichever is later.
* Ongoing Grade >= 2 sensory or motor neuropathy
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, granulomatosis with polyangiitis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions: Patients with a history of autoimmune-mediated hypothyroidism who are on thyroid replacement hormone are eligible for the study. Patients with controlled Type 1 diabetes mellitus are eligible for the study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met: Rash must cover < 10% of body surface area.
* Pharmacologically uncompensated, symptomatic hypothyroidism
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Prior allogeneic stem cell or solid organ transplantation
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication are eligible for the study after Medical Monitor confirmation has been obtained. Patients who received mineralocorticoids, inhaled or low-dose systemic corticosteroids for COPD or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the cabozantinib formulation
* History of severe hypersensitivity to docetaxel or to other drugs formulated with polysorbate 80
* Concomitant anticoagulation with coumarin agents, direct thrombin inhibitor dabigatran, direct factor Xa inhibitor betrixaban, or platelet inhibitors
* History of risk factors for torsades de pointes
* Corrected QT interval corrected through use of Fridericia's formula (QTcF) > 480 ms per ECG within 14 days before initiation of study treatment
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal antihypertensive treatment
* Tumors invading the GI-tract, active peptic ulcer disease, acute pancreatitis, acute obstruction of the pancreatic or biliary duct, appendicitis, cholangitis, cholecystitis, diverticulitis, gastric outlet obstruction, or inflammatory bowel disease
* Abdominal fistula, bowel obstruction, GI perforation, or intra-abdominal abscess within 6 months before initiation of study treatment
* Known cavitating pulmonary lesion(s) or known endobronchial disease manifestation
* Lesions invading major pulmonary blood vessels
* Clinically significant hematuria, hematemesis, hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, coagulopathy, or other history of significant bleeding within 3 months before initiation of study treatment
* Serious non-healing wound/ulcer/bone fracture
* Malabsorption syndrome
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption are also excluded.
* Requirement for hemodialysis or peritoneal dialysis
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (92):
- United States (12):
  - Stanford University, Palo Alto, California
  - Kaiser Permanente - San Diego, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Regional Cancer Care Associates, Bethesda, Maryland
  - Minnesota Oncology Hematology, Saint Paul, Minnesota
  - Consultants in Medical Oncology and Hematology, Broomall, Pennsylvania
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
  - Oncology and Hematology Associates of Southwest Virginia, Inc.,-Blacksburg, Blacksburg, Virginia
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Townsville Hospital, Townsville, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Hospital Olivia Newton John Cancer Centre, Heidelberg, Victoria
  - Affinity Oncology, Nedlands, Western Australia
- Austria (5):
  - Lkh-Univ. Klinikum Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
  - Lhk Feldkirch, Rankweil
  - Lkh Salzburg - Univ. Klinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires St-Luc, Brussels
  - Clinique Ste-Elisabeth, Namur
- France (6):
  - CHU Angers,Service de Pneumologie, Angers
  - CHU de Grenoble, Grenoble
  - Hopital Dupuytren, Limoges
  - Hôpital Saint Joseph, Marseille
  - Centre Regional de Lutte contre le Cancer Val d Aurelle - Paul Lamarque, Montpellier
  - Hopital Tenon, Paris
- Germany (6):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Klinikum Koeln-Merheim, Cologne
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - KRH Klinikum Siloah-Oststadt-Heidehaus, Hanover
  - Universitaetsklinikum Giessen und Marburg, Marburg
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
- Greece (4):
  - Uoa Sotiria Hospital, Athens
  - Henri Dunant Hospital, Athens
  - Univ General Hosp Heraklion, Heraklion
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
- Italy (11):
  - Ospedale Vito Fazzi, Lecce, Apulia
  - AORN Ospedali dei Colli Ospedale Monaldi, Napoli, Campania
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Ospedale Provinciale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Policlinico Umberto I, Oncologia B, Rome, Lazio
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Instituto Europeo di Oncologia, Milan, Lombardy
  - A.O.U Careggi, Florence, Tuscany
- Japan (5):
  - Hyogo Cancer Center, Hyōgo
  - Sendai Kousei Hospital, Miyagi
  - Osaka International Cancer Institute, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (5):
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - SP ZOZ Wojewódzki Szpital Specjalistyczny nr 4, Bytom
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice, Gliwice
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
- Portugal (4):
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - IPO do Porto, Porto
  - CHVNG/E_Unidade 1, Vila Nova de Gaia
- Russia (4):
  - MEDSI Clinical Hospital on Pyatnitsky Highway, Moscow, Moscow Oblast
  - GBUZ Leningradskaya state clinical hospital, Saint Petersburg, Sankt-Peterburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
- South Korea (12):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - St. Vincent's Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Samsung Changwon Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Institut Catala d Oncologia Hospital Duran i Reynals, L'Hospitalet de LLobegat
  - Hospital Universitario La Paz, Madrid
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (5):
  - Addenbrookes Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts & London School of Med, London
  - University College London Hospital, London
  - Chelsea & Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Neal J, Pavlakis N, Kim SW, Goto Y, Lim SM, Mountzios G, Fountzilas E, Mochalova A, Christoph DC, Bearz A, Quantin X, Palmero R, Antic V, Chun E, Edubilli TR, Lin YC, Huseni M, Ballinger M, Graupner V, Curran D, Vervaet P, Newsom-Davis T. CONTACT-01: A Randomized Phase III Trial of Atezolizumab + Cabozantinib Versus Docetaxel for Metastatic Non-Small Cell Lung Cancer After a Checkpoint Inhibitor and Chemotherapy. J Clin Oncol. 2024 Jul 10;42(20):2393-2403. doi: 10.1200/JCO.23.02166. Epub 2024 Mar 29. PMID 38552197
- [Derived] Xing P, Wang M, Zhao J, Zhong W, Chi Y, Xu Z, Li J. Study protocol: A single-arm, multicenter, phase II trial of camrelizumab plus apatinib for advanced nonsquamous NSCLC previously treated with first-line immunotherapy. Thorac Cancer. 2021 Oct;12(20):2825-2828. doi: 10.1111/1759-7714.14113. Epub 2021 Aug 18. PMID 34409776
- See also: Related Info — https://forpatients.roche.com/en/trials/cancer/lung-cancer/study-of-atezolizumab-in-combination-with-cabozantinib--77103.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 366 participants with metastatic non-small cell lung cancer (NSCLC) previously treated with anti-programmed death ligand 1/programmed cell death protein 1 (PD-L1/PD-1) antibody and platinum-containing chemotherapy took part in the study at 97 investigative sites across 15 countries from 01 October 2020 to 17 January 2025.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either docetaxel monotherapy or atezolizumab & cabozantinib combination therapy. A total of 14 participants did not receive any study treatment and were therefore excluded from the safety analysis.
Groups:
- Docetaxel Monotherapy: Participants received docetaxel, 75 milligrams per square meter (mg/m^2), intravenously (IV) on Day 1 of each 21-day cycle until unacceptable toxicity or disease progression (PD) or loss of clinical benefit as determined by the investigator.
- Atezolizumab + Cabozantinib: Participants received atezolizumab, 1200 milligrams (mg), IV, on Day 1 of each 21-day cycle along with cabozantinib, 40 mg, orally, given once a day (QD) on Days 1-21 of each cycle until unacceptable toxicity, PD, or loss of clinical benefit as determined by the investigator.
Period: Overall Study
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Started | 180 | 186
Safety-evaluable Population (Safety-evaluable population included all randomized participants who had received any amount of study drug, with participants grouped according to the actual treatment received.) | 167 | 185
Completed | 0 | 0
Not Completed | 180 | 186
Not completed — Withdrawal by Subject | 29 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Reason Not Specified | 0 | 2
Not completed — Death | 131 | 147
Not completed — Lost to Follow-up | 0 | 3
Not completed — Study Terminated by Sponsor | 20 | 29

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants, whether or not the participant received the assigned treatment.
Groups:
- Docetaxel Monotherapy: Participants received docetaxel, 75 mg/m^2, IV on Day 1 of each 21-day cycle until unacceptable toxicity or PD or loss of clinical benefit as determined by the investigator.
- Atezolizumab + Cabozantinib: Participants received atezolizumab, 1200 mg, IV, on Day 1 of each 21-day cycle along with cabozantinib, 40 mg, orally, given QD on Days 1-21 of each cycle until unacceptable toxicity, PD, or loss of clinical benefit as determined by the investigator.
- Total: Total of all reporting groups
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib | Total
Number analyzed (Participants) | 180 | 186 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.4) | 63.8 (9.5) | 64.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 105
  Male | 127 | 134 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 53 | 41 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 111 | 130 | 241
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 158 | 164 | 322
  Not Stated | 12 | 15 | 27
  Unknown | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause. Participants alive at the time of the analysis were censored at the date when they were last known to be alive as documented by the investigator. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 24 months
Population: The ITT population included all randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
months | 10.5 [8.6 to 13.0] | 10.7 [8.8 to 12.3]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Test type: Superiority — Stratified Analysis: Stratification factors include histology, and prior NSCLC treatment regimens; p = 0.3668, Log Rank; Hazard Ratio (HR) = 0.884, 95% CI 2-sided [0.676 to 1.156] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified Analysis; Test type: Superiority; p = 0.4709, Log Rank; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.696 to 1.182] — Hazard ratio was estimated by Cox regression model

2. Secondary Outcome: Progression-Free Survival (PFS) as Determined by Investigator
Description: PFS was defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1), or death from any cause (whichever occurred first). PD was defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters of the target lesions recorded since the treatment started, including screening, or the appearance of one or more new lesions. In addition, the sum of diameters also demonstrated an absolute increase of ≥ 5 millimeters (mm). Participants who were alive and did not experience PD at the time of analysis, were censored on the date of last tumor assessment. Participants with no post-baseline tumor assessment were censored at the date of randomization. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 24 months
Population: The ITT population included all randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
months | 4.0 [3.1 to 4.4] | 4.6 [4.1 to 5.6]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Stratified Analysis; Stratification factors include histology, and prior NSCLC treatment regimens; Test type: Superiority; p = 0.0079, Log Rank; Hazard Ratio (HR) = 0.735, 95% CI 2-sided [0.585 to 0.923] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified analysis; Test type: Superiority; p = 0.0061, Log Rank; Hazard Ratio (HR) = 0.731, 95% CI 2-sided [0.583 to 0.915] — Hazard ratio was estimated by Cox regression model

3. Secondary Outcome: Confirmed Objective Response Rate (ORR) as Determined by Investigator
Description: Confirmed ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to RECIST v1.1. CR= disappearance of all target lesions. In addition, any pathological lymph nodes must have a reduction in short axis to < 10 mm. PR= at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters. 95% CIs for rates were constructed using the Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Up to approximately 24 months
Population: The ITT population included all randomized participants, whether or not the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
percentage of participants | 13.3 [8.73 to 19.19] | 11.8 [7.56 to 17.36]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Stratified analysis; stratification factors- histology, prior NSCLC treatment regimens; Test type: Superiority; p = 0.6846, Cochran-Mantel-Haenszel; Difference in Response Rates = -1.51, 95% CI 2-sided [-8.85 to 5.84] — 95% CIs was computed using the Wald method
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Stratified analysis; stratification factors- histology, prior NSCLC treatment regimens; Test type: Superiority; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.47 to 1.63] — Odds ratios were estimated by logistic regression. 95% CIs was computed using the Wald method
Statistical Analysis 3: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified Analysis; Test type: Superiority; p = 0.7216, Chi-squared, Corrected; Difference in Response Rates = -1.51, 95% CI 2-sided [-8.85 to 5.84] — 95% CIs was computed using the Wald method
Statistical Analysis 4: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified Analysis; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.47 to 1.62] — Odds ratios were estimated by logistic regression. 95% CIs was computed using the Wald method

4. Secondary Outcome: Duration of Response (DOR) as Determined by Investigator
Description: DOR for participants with confirmed ORR=time from first documented objective response to PD, as determined by investigator per RECIST v1.1, or death from any cause (whichever occurred first). PD=≥ 20% increase in sum of longest diameters of target lesions, taking as reference smallest sum of longest diameters of target lesions recorded since treatment started, including screening, or appearance of new lesions. In addition, sum of diameters also demonstrated an absolute increase of ≥ 5 mm. Confirmed ORR=percentage of participants with a CR or PR on two consecutive occasions ≥4 weeks apart, as determined by investigator per RECIST v1.1. CR= disappearance of all target lesions. PR=≥ 30% decrease in sum of diameters of all target lesions. Participants who had not progressed and who did not die at the time of analysis were censored at the time of last tumor assessment date. Kaplan-Meier method was used to estimate median. 95% CI for median was computed using Brookmeyer and Crowley method.
Time Frame: Up to approximately 24 months
Population: Participants in the ITT population who had a confirmed objective response (CR or PR) as determined by the investigator per RECIST v1.1 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 24 | 22
months | 4.30 [3.29 to 5.62] | 5.55 [3.12 to 10.25]

5. Secondary Outcome: Time to Confirmed Deterioration (TTCD) in Patient-reported Physical Functioning (PF)
Description: TTCD analyses was performed for patient-reported PF (items 1 to 5) of European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30). The PF was measured on 4-point scale (1='Not at all' to 4='Very much'). TTCD for PF was defined as time from date of randomization to first confirmed clinically meaningful decrease from baseline in PF score held for at least 2 consecutive assessments or initial clinically meaningful decrease from baseline followed by death from any cause within 21 days or until next tumor assessment, whichever occurs first. A score change of ≥ of 10-point on EORTC QLQ-C30 PF scale was determined as being clinically meaningful. Scores were averaged, transformed to 0-100 scale; where higher score represented high/healthy level of functioning. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 24 months
Population: The ITT population included all randomized participants, whether or not the participant received the assigned treatment. Participants without a confirmed deterioration at the time of analysis were censored at the last time they were known to have not deteriorated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
months | 5.6 [4.0 to NA] — Upper limit of 95% confidence interval (CI) was not estimable as there were not enough events after the median estimate to satisfy constraints required to calculate the upper limit of interval. | 7.7 [4.8 to 14.7]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Stratified Analysis: Stratification factors include histology, and prior NSCLC treatment regimens; Test type: Superiority; p = 0.2700, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.59 to 1.16] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified Analysis; Test type: Superiority; p = 0.3031, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.60 to 1.17] — Hazard ratio was estimated by Cox regression model

6. Secondary Outcome: TTCD in Patient-reported Global Health Status (GHS)
Description: TTCD analyses was performed for GHS and quality of life (QoL) (items 29 and 30) of EORTC QLQ-C30. GHS/ QoL items were scored on a 7-point scale that ranges from "very poor" to "excellent." TTCD for GHS/QoL was defined as the time from the date of randomization to the first confirmed clinically meaningful decrease from baseline in GHS/QoL score held for at least two consecutive assessments or an initial clinically meaningful decrease from baseline followed by death from any cause within 21 days or until the next tumor assessment, whichever occurs first. A score change of ≥ 10-point on the EORTC QLQ-C30 GHS/QoL scale was determined as being clinically meaningful. Scores were averaged, transformed to 0-100 scale; where higher score for GHS/QoL= better health-related QoL. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 24 months
Population: Participants without a confirmed deterioration at the time of analysis were censored at the last time they were known to have not deteriorated. The ITT population included all randomized participants, whether or not the participant received the assigned treatment. Only responders were analysed in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
months | 14.1 [6.3 to NA] — Upper limit of 95% confidence interval (CI) was not estimable as there were not enough events after the median estimate to satisfy constraints required to calculate the upper limit of interval. | 8.1 [5.6 to 14.5]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Stratification factors include histology, and prior NSCLC treatment regimens; Test type: Superiority; p = 0.2408, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.86 to 1.79] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; Unstratified Analysis; Test type: Superiority; p = 0.1992, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.88 to 1.81] — Hazard ratio was estimated by Cox regression model

7. Secondary Outcome: PFS Rates Assessed by Investigator
Description: PFS rates were defined as the percentage of participants alive and without PD as assessed by the investigator according to RECIST v1.1 at 6 months and 1 year after randomization. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints, including baseline. In addition, the sum of diameters also demonstrated an absolute increase of ≥ 5 mm. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley. Percentages have been rounded off.
Time Frame: 6 months and 1 year
Population: The ITT population included all randomized participants, whether or not the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
percentage of participants
  At 6 months | 23.66 [16.98 to 30.33] | 39.51 [32.42 to 46.59]
  At 1 year | 8.38 [3.95 to 12.80] | 14.70 [9.43 to 19.97]
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; At 6 months; Test type: Superiority; p = 0.0014, z-test; Difference in Event Free Rate = 15.85, 95% CI 2-sided [6.12 to 25.59] — The 95% CI for the difference in PFS rates were estimated using the normal approximation method, with standard errors computed using the Greenwood method
Statistical Analysis 2: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; At 1 year; Test type: Superiority; p = 0.0719, z-test; Difference in Event Free Rate = 6.32, 95% CI 2-sided [-0.56 to 13.21] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: OS Rates
Description: OS rates were defined as the percentage of participants who were alive at 1 and 2 years. Participants alive at the time of the analysis were censored at the date when they were last known to be alive as documented by the investigator. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley. Percentages have been rounded off.
Time Frame: 1 and 2 years
Population: The ITT population is defined as all randomized participants, whether or not the participant received the assigned treatment. Participants alive at the time of the analysis were censored at the date when they were last known to be alive as documented by the investigator. At the time of the analysis, there were no participants with 24 months or more of survival follow-up, therefore, survival rate at the 2-year timepoint was not estimable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 180 | 186
percentage of participants
  1 year | 44.12 [36.20 to 52.05] | 43.27 [35.97 to 50.57]
  2 years | NA [NA to NA] — Participants alive at the time of the analysis of the 2-year time point were censored at the date when they were last known to be alive as documented by the investigator. There were no participants with 24 months or more of survival follow-up, therefore, survival rate at the 2-year time point was not estimable. | NA [NA to NA] — Participants alive at the time of the analysis of the 2-year time point were censored at the date when they were last known to be alive as documented by the investigator. There were no participants with 24 months or more of survival follow-up, therefore, survival rate at the 2-year time point was not estimable.
Statistical Analysis 1: Comparison: Docetaxel Monotherapy vs Atezolizumab + Cabozantinib; At 1 year; Test type: Superiority; p = 0.8767, z-test; Difference in Event Free Rate = -0.85, 95% CI 2-sided [-11.63 to 9.92] — The 95% CI for the difference in OS rates were estimated using the normal approximation method, with standard errors computed using the Greenwood method

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following: unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product; any new disease or exacerbation of an existing disease; recurrence of an intermittent medical condition not present at baseline; any deterioration in a laboratory value or other clinical test; AEs related to a protocol-mandated intervention. AEs were assessed using National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v5.0). Percentages have been rounded off.
Time Frame: Up to approximately 41.4 months
Population: Safety-evaluable population included all randomized participants who had received any amount of study drug, with participants grouped according to the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 167 | 185
percentage of participants | 94.0 | 98.4

10. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, 8, 12 and 16 (Cycle= 21 days)
Population: Pharmacokinetic (PK)-evaluable population for atezolizumab included all participants who had received any dose of atezolizumab and who had evaluable PK samples. Number analyzed is the number of participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/ml)
Arm/Group | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 185
microgram/milliliter (μg/ml)
  Cycle 1 Day 1: number analyzed (Participants) | 146
  Cycle 1 Day 1 | NA (NA) — The data was not evaluable as all samples were below limit of quantitation (BLQ)
  Cycle 2 Day 1: number analyzed (Participants) | 162
  Cycle 2 Day 1 | 96.8 (48.1)
  Cycle 3 Day 1: number analyzed (Participants) | 140
  Cycle 3 Day 1 | 124 (104.4)
  Cycle 4 Day 1: number analyzed (Participants) | 130
  Cycle 4 Day 1 | 167 (47.7)
  Cycle 8 Day 1: number analyzed (Participants) | 70
  Cycle 8 Day 1 | 194 (62.4)
  Cycle 12 Day 1: number analyzed (Participants) | 52
  Cycle 12 Day 1 | 233 (44.7)
  Cycle 16 Day 1: number analyzed (Participants) | 40
  Cycle 16 Day 1 | 209 (56.1)

11. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: 30 minutes (min) postdose on Day 1 of Cycle 1 (Cycle= 21 days)
Population: PK-evaluable population included all participants who had received any dose of atezolizumab and who had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 185
μg/mL | 450 (34.0)

12. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Cabozantinib
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, and 5 (Cycle= 21 days)
Population: PK-evaluable population included all participants who had received any dose of cabozantinib and who had evaluable PK samples. Number analyzed is the number of participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 185
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 173
  Cycle 1 Day 1 | NA (NA) — The data was not evaluable as all samples were Below Limit of Quantitation (BLQ)
  Cycle 2 Day 1: number analyzed (Participants) | 163
  Cycle 2 Day 1 | 0.746 (111.7)
  Cycle 3 Day 1: number analyzed (Participants) | 138
  Cycle 3 Day 1 | 0.418 (640.7)
  Cycle 4 Day 1: number analyzed (Participants) | 131
  Cycle 4 Day 1 | 0.469 (234.4)
  Cycle 5 Day 1: number analyzed (Participants) | 110
  Cycle 5 Day 1 | 0.303 (402.3)

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Cabozantinib
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, and 5 (Cycle= 21 days)
Population: Cmax was not collected for this outcome measure because PK of cabozantinib was well characterized through the cabozantinib development for mono- therapy. An established population PK model for cabozantinib is available for the PK data from NCT04471428 (study GO41892). The PK data collected in the current study is sufficient for the population PK model to characterize the exposure of cabozantinib in this study.
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Participants were considered to be ADA positive if they were ADA negative or had missing data at baseline but developed an ADA response following study drug exposure (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples was at least 0.60 titer unit greater than the titer of the baseline sample (treatment-enhanced ADA response). The total number of participants who developed ADAs to atezolizumab was determined by summing the ADA-positive participants across all timepoints.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3, 4, 8, 12, 16 and post-treatment follow-up (≤ 30 days after final dose) (Cycle= 21 days)
Population: Safety-evaluable population included all randomized participants who had received any amount of study drug, with participants grouped according to the actual treatment received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 177
Participants
  ADA Prevalence at Baseline | 2
  ADA Incidence after treatment: number analyzed (Participants) | 173
  ADA Incidence after treatment | 37

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 44.6 months SAE and other AEs: Up to 41.4 months
Description: Safety-evaluable population which included all randomized participants who had received any amount of study drug. A total of 14 participants did not receive any study treatment and were therefore excluded from the safety analysis. All-cause mortality reported for deaths that occurred during study based on ITT population.
Arm/Group | Docetaxel Monotherapy | Atezolizumab + Cabozantinib
All-Cause Mortality (participants affected / at risk) | 131/180 | 147/186
Serious Adverse Events (participants affected / at risk) | 58/167 | 76/185
Other Adverse Events (participants affected / at risk) | 148/167 | 173/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel Monotherapy (N=167) | Atezolizumab + Cabozantinib (N=185)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pneumopericardium (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (3) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (2)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 5 (6)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 10 (10)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (2)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel Monotherapy (N=167) | Atezolizumab + Cabozantinib (N=185)
Anaemia (Blood and lymphatic system disorders) | 38 (47) | 24 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 17 (20)
Hypothyroidism (Endocrine disorders) | 0 (0) | 30 (32)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 21 (27)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 11 (12)
Constipation (Gastrointestinal disorders) | 17 (17) | 31 (35)
Diarrhoea (Gastrointestinal disorders) | 38 (62) | 83 (134)
Nausea (Gastrointestinal disorders) | 29 (42) | 47 (56)
Stomatitis (Gastrointestinal disorders) | 13 (14) | 28 (30)
Vomiting (Gastrointestinal disorders) | 11 (14) | 29 (36)
Asthenia (General disorders) | 40 (45) | 43 (53)
Fatigue (General disorders) | 44 (48) | 42 (48)
Malaise (General disorders) | 9 (9) | 5 (5)
Mucosal inflammation (General disorders) | 9 (10) | 11 (17)
Oedema peripheral (General disorders) | 12 (15) | 8 (8)
Pyrexia (General disorders) | 12 (12) | 20 (21)
COVID-19 (Infections and infestations) | 4 (4) | 14 (15)
Alanine aminotransferase increased (Investigations) | 7 (7) | 36 (53)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 31 (42)
Neutrophil count decreased (Investigations) | 12 (19) | 8 (17)
Platelet count decreased (Investigations) | 0 (0) | 15 (27)
Weight decreased (Investigations) | 6 (7) | 30 (30)
Decreased appetite (Metabolism and nutrition disorders) | 28 (31) | 59 (64)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (16) | 20 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 20 (35)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9) | 15 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 23 (29)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 12 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (23) | 26 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 18 (20)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (23) | 11 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 12 (15)
Dizziness (Nervous system disorders) | 5 (5) | 14 (15)
Dysgeusia (Nervous system disorders) | 10 (14) | 20 (24)
Headache (Nervous system disorders) | 14 (18) | 14 (16)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7) | 17 (18)
Proteinuria (Renal and urinary disorders) | 3 (3) | 22 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 20 (25)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 27 (29)
Alopecia (Skin and subcutaneous tissue disorders) | 40 (40) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 11 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 40 (54)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 15 (19)
Rash (Skin and subcutaneous tissue disorders) | 13 (14) | 17 (20)
Hypertension (Vascular disorders) | 2 (3) | 17 (25)
Amylase increased (Investigations) | 2 (2) | 10 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT04471428/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT04471428/SAP_001.pdf